CLINICAL TRIAL: NCT02688699
Title: Italian Multicenter Prospective Randomized Trial to Compare Additive Hemostatic Efficacy of EndoClot System to Prevent Bleeding After Endoscopic Mucosal Resection or Endoscopic Submucosal Dissection of Lesions in the Gastrointestinal Tract
Brief Title: Additive Hemostatic Efficacy of EndoClot After EMR or ESD in the Gastrointestinal Tract
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Alberto Arezzo, Associate Professor of Surgery, MD, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12243648
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Colonic Polyp; Colonic Neoplasms; Colonic Dysplasia
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EndoClot (Experimental): spraying of Endoclot powder after EMR or ESD
  Interventions: Procedure: EndoClot
- control (No Intervention)

INTERVENTIONS:
Procedure: EndoClot — All patients enrolled and submitted to EMR or ESD in several units of Italian endoscopy will be divided into two different groups: in a first group will be included patients at the endoscopic end of which will be applied EndoClotTM based on the lesion removed in addition to the treatment Standard (drug injection, electrocoagulation, metal clips). The second group, on the other hand, includes patients in whom EndoClotTM will not be used.
  Before the end of the procedure neither the endoscopist nor the patient will know the group because the group to which the patient is assigned will be written in a sealed envelope that will be opened only at the end of the procedure before the endoscope extraction: The use of EndoClotTM will depend on the group to which the patient belongs.
  Arms: EndoClot

SUMMARY:
The investigators want to verify in a randomised trial, the effectiveness of EndoClotTM in preventing post-procedural bleeding after EMR (Endoscopic Mucosal Resection) or ESD (Endoscopic Submucosal Dissection) for sessile lesions >20 mm in the right colon

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* lesions suitable for EMR or ESD
* > 20 mm
* site in the right colon

Exclusion Criteria:

* Severe cardiovascular pathologies
* Liver and Urinary dysfunctions
* Hematologic diseases
* Pregnancy and breast feeding
* impossible follow-up
* platelet and coagulation disorders (PLT < 50 x 109/L, INR > 2)
* Sensitivity or allergy to the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
effectiveness of EndoClotTM in preventing post-procedural bleeding | 14 days
  The investigators want to verify in a randomised trial, the effectiveness of EndoClotTM in preventing post-procedural bleeding after EMR (Endoscopic Mucosal Resection) or ESD (Endoscopic Submucosal Dissection) for sessile lesions >20 mm in the right colon